CLINICAL TRIAL: NCT01134406
Title: A Prospective, Multi-center, Randomized, Double-blind Feasibility Study to Evaluate the Safety and Performance of Hydros Joint Therapy and Hydros-TA Joint Therapy for Management of Pain Associated With Osteoarthritis in the Knee
Brief Title: Hydros Joint Therapy and Hydros-TA Joint Therapy for Pain Associated With Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carbylan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COR 1.0
Record Dates: First submitted 2010-05-05; First posted 2010-06-02 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydros Joint Therapy (Experimental): Experimental viscosupplement.
  Interventions: Device: Hydros Joint Therapy
- Hydros-TA Joint Therapy (Experimental): Experimental viscosupplement.
  Interventions: Device: Hydros-TA Joint Therapy
- Synvisc-One (Active Comparator): Commercial control.
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: Hydros Joint Therapy — Single intra-articular injection.
  Other Names: Hydros
  Arms: Hydros Joint Therapy
Device: Hydros-TA Joint Therapy — Single intra-articular injection
  Other Names: Hydros-TA
  Arms: Hydros-TA Joint Therapy
Device: Synvisc-One — Single intra-articular injection.
  Other Names: Hylan G-F 20
  Arms: Synvisc-One

SUMMARY:
The purpose of this study is to evaluate the safety and performance of Hydros Joint Therapy (Hydros) and Hydros-TA Joint Therapy (Hydros-TA) for treatment of pain from osteoarthritis of the knee, in patients who have failed to respond adequately to conservative non-pharmacologic therapy and simple analgesics.

DETAILED DESCRIPTION:
The objective of the study is to evaluate Hydros and Hydros-TA treated subject for reduction of osteoarthritis symptoms, compared to a commercial control, as assessed by the WOMAC Osteoarthritis Index.

The WOMAC Osteoarthritis Index is a validated assessment instrument that is self-administered and designed to subjectively elicit patient symptoms of osteoarthritis in the knee in the areas of pain, stiffness, and physical function. The WOMAC Osteoarthritis Index with its Pain Subscale has been used extensively as an effectiveness endpoint in clinical trials of viscosupplements.

ELIGIBILITY:
Inclusion Criteria:

- Osteoarthritis grade 2 or 3 in one knee using Kellgren-Lawrence Grading for OA radiologically and verified within the prior 6 months.

Exclusion Criteria:

* Secondary OA resulting from rheumatoid arthritis, chondrocalcinosis, osteonecrosis, chronic fibromyalgia or other autoimmune disease.
* Generalized symptomatic OA in lower extremity joints other than the knees.
* Active infection in either knee joint or adjacent tissues.
* Any contraindications for intra-articular injection or aspiration.
* Knee surgery or trauma within 3 months prior to enrollment.
* Intra-articular steroid injection in the knee and/or use of systemic (oral) corticosteroids within 3 months prior to enrollment.
* Intra-articular hyaluronan injection in the treatment knee within 6 months prior to enrollment.
* Body Mass Index (BMI) greater than 35.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
WOMAC VAS Pain over 26 weeks | 26 weeks post treatment

SECONDARY OUTCOMES:
WOMAC VAS Stiffness and Function over 26 weeks | 26 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Research, London, Ontario, Canada

REFERENCES:
- [Derived] Petrella RJ, Emans PJ, Alleyne J, Dellaert F, Gill DP, Maroney M. Safety and performance of Hydros and Hydros-TA for knee osteoarthritis: a prospective, multicenter, randomized, double-blind feasibility trial. BMC Musculoskelet Disord. 2015 Mar 18;16:57. doi: 10.1186/s12891-015-0513-6. PMID 25887932